CLINICAL TRIAL: NCT01255449
Title: Predictive Value of Within-breath Respiratory Input Impedance in the Early Diagnosis of Obliterative Bronchiolitis After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Respiratory Impedance and Obliterative Bronchiolitis
Acronym: FOT-BOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Barisione, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FOT-BOS-01
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-12

CONDITIONS: Hematopoietic Stem Cell Transplantation; Obliterative Bronchiolitis
Keywords: Forced oscillation technique; Respiratory input impedance; Allogeneic hematopoietic stem cell transplantation; Obliterative bronchiolitis
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- albuterol (Experimental): Twenty-six consecutive patients undergoing allogeneic HSCT for hematological malignancies were studied. All patients were in stable clinical conditions at the time of study. All patients received a myeloablative conditioning regimen either including or not including total body irradiation. Spirometry, lung volumes, FOT and lung CT scan were obtained before the start of conditioning treatment and, approximately, two months after HSCT. On each study day, all the above measurements were taken before and 30 min after inhaling four consecutive albuterol doses, of 100 mcg each, through a valved-holding chamber. DLco was measured only after bronchodilator inhalation.
  Interventions: Drug: albuterol

INTERVENTIONS:
Drug: albuterol — 400 mcg by inhalation
  Other Names: Broncovaleas pressurized solution

SUMMARY:
The aim of the present study will be to test the hypothesis that changes in within-breath total respiratory input impedance (Zrs) may provide an early evidence of obliterative bronchiolitis after allogeneic hematopoietic stem cell transplantation (HSCT). Before and after HSCT, Zrs will be measured by a modified forced oscillation technique (FOT) during spontaneous breathing both at baseline and 30 min after albuterol inhalation . Such technique may be particularly sensitive to small changes in lung mechanics observed in the early stages of peripheral airflow obstruction.

DETAILED DESCRIPTION:
1.0 INTRODUCTION

* Shortly after the introduction of allogeneic HSCT in clinical practice, it was recognized that standard pulmonary function tests (PFTs) are sensitive enough to detect HSCT-related respiratory complications [PMID: 2661259; PIMD: 8823260]. Accordingly, the finding of a progressive obstructive abnormality of new onset was considered as the functional hallmark of obliterative bronchiolitis (OB) [PMID: 16338616; PMID: 19896545]. As a result, routinely performed spirometry has been proposed as a non-invasive tool to monitor the risk of OB in HSCT population [PMID: 17470622]. Yet, due to a peripheral airway involvement in OB, the sensitivity of conventional PFTs for early detection of OB is low [PMID: 2298060]. For instance, it does not exceed 75% in lung-transplanted population as the decrease of forced expiratory volume in 1 s (FEV1) may occur at a stage when the process is already irreversible and potentially life-threatening [PMID: 9246138].

2.0 EXPERIMENTAL HYPOTHESIS

* Because the branching pattern of the bronchial tree results in an increasingly large number of small airways with a luminal diameter of less than 2 mm in peripheral generations, these airways contribute little to total pulmonary resistance [PMID: 5442364; PMID: 651978]. Intuitively, a large proportion of small airways may be damaged or obliterated without impairing any of the conventional PFTs. In this regard, a previous study [PMID: 12186817] pointed out that indexes of ventilation distribution may provide an early evidence of OB after lung transplantation. In particular, some authors [PMID: 12186817] have found that tests of ventilation distribution invariably deteriorated about 1 yr before a 20% decrease in FEV1 was apparent. Previous studies [PMID: 970731; PMID: 507525] showed that total respiratory input impedance (Zrs), measured by a forced oscillation technique (FOT) during spontaneous breathing, may be particularly sensitive to small changes in lung mechanics observed in the early stages of smoking-related airflow obstruction. Subsequently, it was developed a modified FOT to identify within-breath differences in Zrs, with values of Zrs representing the sum of respiratory system resistance (Rrs) and reactance (Xrs), the latter being the imaginary part of the former [PMID: 14979497; PMID: 19164347]. This method allows the assessment of more breaths and adds a potential quantitative evaluation of instantaneous inspiratory and expiratory Rrs and Xrs before and after external interventions such as a deep inspiration, bronchodilator drugs, etc. Although these effects can be identified when within-breath analysis is performed [PMID: 14979497], most published reports of oscillatory mechanics on chronic obstructive pulmonary disease (COPD) only report total respiratory cycle data [PMID: 1519830; PMID: 10489847].

3.0 STUDY RATIONALE

* The aim of the present study will be to test the hypotheses that:

  1. post-HSCT changes in within-breath Rrs and Xrs may provide an earlier evidence of OB than standard PFTs. Indeed, the obliteration of terminal bronchioles, observed in up to 48% of OB patients following HSCT [PMID: 17470622], could make the real part of Zrs abnormally high [PMID: 5653219] and ventilation more heterogeneous;
  2. post-HSCT changes of airway responsiveness to acute bronchoactive interventions such as a deep inspiration to total lung capacity and/or a bronchodilator drug (i.e., albuterol) may be detected by our modified FOT. We speculate that these changes may represent an early sign of OB. Although a previous study from our group failed to find an increase in airway responsiveness after HSCT without pulmonary complications [PMID: 18684842], we have recently shown that airway smooth muscle tone may play an active role in the airflow obstruction of OB [PMID: 20724742].

4.0 STUDY DESIGN

* Before and at regular intervals (2-4 wk onward) after HSCT, patients will attend our laboratory and perform all PFTs measurements in the same order. Firstly, the patient will breathe spontaneously through the modified FOT system for 5 min and then, without disconnecting from the apparatus, perform an inspiratory capacity maneuver and soon after resume spontaneous breathing for the next 2 min. Subsequently, spirometry, transmural total body plethysmography and CO diffusing capacity of the lung (standard PFTs) will be taken in triplicate. Thirty minutes after inhaling four separate doses of 100 μg of albuterol, the modified FOT measurements and standard PFTs will be repeated anew.

ELIGIBILITY:
Inclusion Criteria:

* consecutive, clinically-stable, outpatients undergoing allogeneic HSCT (sourcing from bone marrow) for hematological malignancies
* values of standard PFTs within normal range before HSCT
* good collaboration during the maneuvers

Exclusion Criteria:

* patients showing any spirometric and/or volumetric abnormality before HSCT
* poor collaboration and/or coordination during the maneuvers
* any clinically-significant respiratory disease (bronchial asthma, COPD, cystic fibrosis, etc.) before HSCT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barisione, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- U.O. Medicina Preventiva e del Lavoro, Laboratorio di Fisiopatologia Respiratoria, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genova, Italy

REFERENCES:
- [Background] Rodriguez-Roisin R, Roca J, Granena A, Agusti AG, Marin P, Rozman C. Lung function in allogeneic bone marrow transplantation recipients. Eur Respir J. 1989 Apr;2(4):359-65. PMID 2661259
- [Background] Gore EM, Lawton CA, Ash RC, Lipchik RJ. Pulmonary function changes in long-term survivors of bone marrow transplantation. Int J Radiat Oncol Biol Phys. 1996 Aug 1;36(1):67-75. doi: 10.1016/s0360-3016(96)00123-x. PMID 8823260
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Chien JW, Duncan S, Williams KM, Pavletic SZ. Bronchiolitis obliterans syndrome after allogeneic hematopoietic stem cell transplantation-an increasingly recognized manifestation of chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2010 Jan;16(1 Suppl):S106-14. doi: 10.1016/j.bbmt.2009.11.002. Epub 2009 Nov 5. PMID 19896545
- [Background] Soubani AO, Uberti JP. Bronchiolitis obliterans following haematopoietic stem cell transplantation. Eur Respir J. 2007 May;29(5):1007-19. doi: 10.1183/09031936.00052806. PMID 17470622
- [Background] Otulana BA, Higenbottam T, Ferrari L, Scott J, Igboaka G, Wallwork J. The use of home spirometry in detecting acute lung rejection and infection following heart-lung transplantation. Chest. 1990 Feb;97(2):353-7. doi: 10.1378/chest.97.2.353. PMID 2298060
- [Background] Van Muylem A, Melot C, Antoine M, Knoop C, Estenne M. Role of pulmonary function in the detection of allograft dysfunction after heart-lung transplantation. Thorax. 1997 Jul;52(7):643-7. doi: 10.1136/thx.52.7.643. PMID 9246138
- [Background] Mead J. The lung's "quiet zone". N Engl J Med. 1970 Jun 4;282(23):1318-9. doi: 10.1056/NEJM197006042822311. No abstract available. PMID 5442364
- [Background] Cosio M, Ghezzo H, Hogg JC, Corbin R, Loveland M, Dosman J, Macklem PT. The relations between structural changes in small airways and pulmonary-function tests. N Engl J Med. 1978 Jun 8;298(23):1277-81. doi: 10.1056/NEJM197806082982303. PMID 651978
- [Background] Estenne M, Hertz MI. Bronchiolitis obliterans after human lung transplantation. Am J Respir Crit Care Med. 2002 Aug 15;166(4):440-4. doi: 10.1164/rccm.200201-003pp. No abstract available. PMID 12186817
- [Background] Kjeldgaard JM, Hyde RW, Speers DM, Reichert WW. Frequency dependence of total respiratory resistance in early airway disease. Am Rev Respir Dis. 1976 Sep;114(3):501-8. doi: 10.1164/arrd.1976.114.3.501. PMID 970731
- [Background] Hayes DA, Pimmel RL, Fullton JM, Bromberg PA. Detection of respiratory mechanical dysfunction by forced random noise impedance parameters. Am Rev Respir Dis. 1979 Nov;120(5):1095-100. doi: 10.1164/arrd.1979.120.5.1095. PMID 507525
- [Background] Dellaca RL, Santus P, Aliverti A, Stevenson N, Centanni S, Macklem PT, Pedotti A, Calverley PM. Detection of expiratory flow limitation in COPD using the forced oscillation technique. Eur Respir J. 2004 Feb;23(2):232-40. doi: 10.1183/09031936.04.00046804. PMID 14979497
- [Background] Dellaca RL, Pompilio PP, Walker PP, Duffy N, Pedotti A, Calverley PM. Effect of bronchodilation on expiratory flow limitation and resting lung mechanics in COPD. Eur Respir J. 2009 Jun;33(6):1329-37. doi: 10.1183/09031936.00139608. Epub 2009 Jan 22. PMID 19164347
- [Background] Chalker RB, Celli BR, Habib RH, Jackson AC. Respiratory input impedance from 4 to 256 Hz in normals and chronic airflow obstruction: comparisons and correlations with spirometry. Am Rev Respir Dis. 1992 Sep;146(3):570-6. doi: 10.1164/ajrccm/146.3.570. PMID 1519830
- [Background] Farre R, Peslin R, Rotger M, Barbera JA, Navajas D. Forced oscillation total respiratory resistance and spontaneous breathing lung resistance in COPD patients. Eur Respir J. 1999 Jul;14(1):172-8. doi: 10.1034/j.1399-3003.1999.14a29.x. PMID 10489847
- [Background] Grimby G, Takishima T, Graham W, Macklem P, Mead J. Frequency dependence of flow resistance in patients with obstructive lung disease. J Clin Invest. 1968 Jun;47(6):1455-65. doi: 10.1172/JCI105837. PMID 5653219
- [Background] Barisione G, Bacigalupo A, Crimi E, Van Lint MT, Lamparelli T, Brusasco V. Changes in lung volumes and airway responsiveness following haematopoietic stem cell transplantation. Eur Respir J. 2008 Dec;32(6):1576-82. doi: 10.1183/09031936.0139807. Epub 2008 Aug 6. PMID 18684842
- [Background] Barisione G, Bacigalupo A, Crimi E, Brusasco V. Acute bronchodilator responsiveness in bronchiolitis obliterans syndrome following hematopoietic stem cell transplantation. Chest. 2011 Mar;139(3):633-639. doi: 10.1378/chest.10-1442. Epub 2010 Aug 19. PMID 20724742
- [Result] Barisione G, Pompilio PP, Bacigalupo A, Brusasco C, Cioe A, Dellaca RL, Lamparelli T, Garlaschi A, Pellegrino R, Brusasco V. Airway distensibility with lung inflation after allogeneic haematopoietic stem-cell transplantation. Respir Physiol Neurobiol. 2012 Oct 15;184(1):80-5. doi: 10.1016/j.resp.2012.07.021. Epub 2012 Aug 8. PMID 22898044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started on 10-Nov-2010 and finished on 15-feb-2012. The recruitment was performed at Pulmonary Function Tests Laboratory of IRCCS AOU San Martino.
Pre-assignment Details: All patients were in stable clinical conditions and none had a history of significant respiratory disease.
Groups:
- Albuterol: On each study day, all lung function measurements were taken before and 30 min after inhaling four consecutive albuterol doses of 100 mcg each, through a valved-holding chamber. Lung diffusing capacity for carbon monoxide was measured only after bronchodilator inhalation.
Period: Overall Study
Arm/Group | Albuterol
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Albuterol: All recruited subjects underwent an acute bronchodilation with albuterol following baseline pulmonary function measurements.
Arm/Group | Albuterol
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Region of Enrollment [Number; unit: participants]
  Italy | 26

OUTCOME MEASURES:

1. Primary Outcome: Airway Distensibility With Lung Inflation After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Description: We studied 26 subjects, 2 weeks before and 2 months after HSCT. Within-breath respiratory system conductance (Grs) at 5, 11 and 19 Hz was measured by forced oscillation technique (FOT) at functional residual capacity (FRC) and total lung capacity (TLC)
Time Frame: 2 weeks before and 2 months after HSCT
Measure: Mean (Standard Deviation); unit: 1/cmH2O*s
Groups:
- Airway Distensibility With Lung Inflation After HSCT: Changes in airway conductance at 5 Hz (Grs5) were related to changes in lung volume (DeltaGrs5/DeltaVL) to estimate airway distensibility
Arm/Group | Airway Distensibility With Lung Inflation After HSCT
Number analyzed (Participants) | 26
1/cmH2O*s | 0.07 (0.10)

2. Secondary Outcome: Post-HSCT Changes in Lung Tissue Density
Description: Changes in lung tissue density were measured by quantitative computed tomography(CT) scan 2 weeks before and 2 months after HSCT
Time Frame: Before and 2 months after HSCT
Population: CT scans, in a format suitable for software analysis, were available in 8 patients only
Measure: Mean (Standard Deviation); unit: g/mL
Groups:
- Post-HSCT Changes in Lung Tissue Density: In eight out of 26 patients, a quantitative CT scan analysis was conducted to measure changes in lung tissue density
Arm/Group | Post-HSCT Changes in Lung Tissue Density
Number analyzed (Participants) | 8
g/mL | 0.03 (0.02)

ADVERSE EVENTS:
Groups:
- Albuterol: All subjects underwent an acute bronchodilation with albuterol by inhaling four consecutive doses (100 mcg each)of the drug through a valved-holding chamber
Arm/Group | Albuterol
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No